CLINICAL TRIAL: NCT03084705
Title: An Interactive, Wearable Device for Measuring and Motivating Hand Use After Stroke
Brief Title: Wearable Device for Motivating Hand Use After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, David Reinkensmeyer, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIH HS# 2017-4119
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manumeter with interactive feedback (Experimental): Study participants will receive an experimental manumeter and interactive feedback from the manumeter to monitor and motivate their upper extremity functional activities.
  Interventions: Device: Manumeter
- Manumeter without interactive feedback (Experimental): Study participants will receive an experimental manumeter but receive no feedback from the manumeter, and will be given the current standard-of-care for increasing upper extremity exercise booklet to perform at home.
  Interventions: Device: Manumeter

INTERVENTIONS:
Device: Manumeter — A manumeter is a first-of-its-kind magnetic sensor to wirelessly detect hand and arm movement in a socially acceptable and easy to don package. The study participants will wear a small magnet as a ring, and a sensing/logging wristband detects changes in the magnetic field as the ring moves; the wristband can detect arm accelerations.

SUMMARY:
The goal of this study is to determine the effectiveness of interactive feedback from a wearable device that senses hand function, the Manumeter, in improving upper extremity function in a pilot, randomized controlled trial with chronic stroke patients

DETAILED DESCRIPTION:
In this randomized controlled trial, the investigators will compare two groups of chronic stroke participants Group 1 of study participants will use the Manumeter with interactive functions to monitor and motivate upper extremity functional activity. Group 2 of study participants will use the Manumeter but receive no feedback and will be given the current standard-of-care, a booklet describing a home exercise program for increasing upper extremity exercise. The investigators hypothesize that study participants who interactively monitor functional activity with the Manumeter will improve their upper extremity function significantly more.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* Experienced one or multiple strokes at least six months previously
* Upper Extremity Fugl-Meyer Score < 60 out of 66
* Absence of moderate to severe upper limb pain (< 3 on the a 10 point visual-analog pain scale)
* Ability to understand the instructions to operate the device

Exclusion Criteria:

* 80 years of age and above
* Implanted pacemaker
* moderate to severe pain in affected arm
* severe tone in affected arm as measured on a standard clinical scale
* language problem that would prevent from properly understanding instructions
* currently pregnant
* difficulty in understanding or complying with the instructions given by the experimenter
* inability to perform the experimental task that will be studied

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Box and Blocks Test (BBT) | 3 months
  To measure unilateral gross manual dexterity

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | 3 months
  To evaluate specific changes in arm function from handling objects differing in size, weight and shape
Fugl-Meyer Motor Assessment (FM) | 3 months
  To assess motor functioning, balance, joint functioning thru performance based movement
Motor Activity Log (MAL) | 3 months
  To evaluate self-reported functional use of the limb
Amount of upper extremity activity | 3 months
  To evaluate the daily amount of upper extremity activity by using the wearable sensor

CONTACTS AND LOCATIONS:
Overall Officials: David Reinkensmeyer, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No